CLINICAL TRIAL: NCT04814875
Title: Phase 1b/2a Study Investigating ATX-101 in Combination With Platinum-based Chemotherapy in Platinum-sensitive, Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: A Study to Evaluate the Combination of ATX-101 and Platinum-based Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: For technical reasons, it was decided by the sponsor to close the ongoing ovarian cancer study, AM ATX101-03, immediately.
Sponsor: THERAPIM PTY LTD (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AM ATX101-03
Record Dates: First submitted 2021-03-04; First posted 2021-03-24 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; High Grade Serious or Endometrioid Carcinoma of the Ovary, Fallopian Tube, or Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 - ACD (Safety) (Experimental): ATX-101 plus carboplatin and pegylated liposomal doxorubicin (ACD)
  Interventions: Drug: ATX-101 + Carboplatin + Pegylated liposomal doxorubicin (ACD)
- Part 2 - ACD (Efficacy) (Experimental): ATX-101 plus carboplatin and pegylated liposomal doxorubicin (ACD)
  Interventions: Drug: ATX-101 + Carboplatin + Pegylated liposomal doxorubicin (ACD)

INTERVENTIONS:
Drug: ATX-101 + Carboplatin + Pegylated liposomal doxorubicin (ACD) — Pegylated liposomal doxorubicin (30 mg/m²) will be administered intravenously on Day 1 of each 28-day cycle; carboplatin (AUC5) will be administered intravenously on Day 1 of each cycle.
  ATX-101 will be administered intravenously on Day 2 of each cycle in three escalation cohorts: 20, 30, and 45 mg/m² according to a 3+3 design.

SUMMARY:
This is a Phase 1b/2a multicenter study, which consists of two parts:

Part 1: the Phase 1b part of the study will investigate the safety of the combination of ATX-101 with carboplatin/pegylated liposomal doxorubicin (ACD). ATX-101 will be administered intravenously in three escalation cohorts: 20, 30, and 45 mg/m² according to a 3+3 design. In the case where 20 mg/m² is not tolerated, the dose can be de-escalated to 15 mg/m².

Part 2: the Phase 2a part of the study will investigate the efficacy and safety of ACD.

ATX-101 will be administered at the dose defined in Part 1 of the study.

Treatment will continue up to six cycles or until disease progression or unacceptable toxicity, participant withdrawal of consent, non-compliance, lost to follow-up, or withdrawal at the Investigators discretion, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age
2. Is not a woman of childbearing potential:

   1. Surgically sterile (i.e., had a bilateral tubal ligation, hysterectomy, salpingectomy, or bilateral oophorectomy at least 6 months prior to Day 1 of the study) or;
   2. Postmenopausal for at least 1 year prior to Day 1 of the study, and have follicle stimulating hormone levels in the postmenopausal range for the study site.
3. Signed written informed consent
4. Histologically confirmed high grade serous or endometrioid carcinoma of the ovary, fallopian tube, or primary peritoneal cancer
5. 1 to 3 prior systemic treatment lines. Prior maintenance therapy with bevacizumab or PARP inhibitors is permitted.
6. Platinum-sensitive carcinoma, defined as disease progression after ≥ 6 months following the most recent platinum-based therapy of the disease
7. Measurable disease on CT/MRI scan according to RECIST 1.1
8. ECOG Performance status 0 to 1
9. Life expectancy of at least 6 months
10. Meet the following laboratory requirements:

    1. Hemoglobin (HGB) ≥ 100 × 109/L
    2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    3. Platelet count ≥ 100 × 109/L
    4. aPTT/PT ≤ 1.5 x ULN
    5. Total bilirubin level ≤ 1.5 × ULN
    6. AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN if liver metastasis present)
    7. Creatinine Clearance > 60 mL/min, as calculated by Cockcroft-Gault formula, or serum creatinine ≤ 1.5 × ULN.

Exclusion Criteria:

1. Have received an anti-cancer/investigational drug within 4 weeks prior to study drug administration
2. Have received a vaccine for COVID-19 within 14 days prior to the first dose of ATX-101 or are scheduled/intend to have a COVID-19 vaccine on Day 1 or during the DLT period (i.e. C1D2 [Day 2] through to C2D2 [Day 30]) of the study
3. Have not recovered from AEs (≥ CTCAE Grade 2 other than alopecia) due to agent(s) administered more than 4 weeks earlier
4. Radiotherapy within 4 weeks prior to study drug administration
5. Major surgery or significant trauma within 28 days (4 weeks) of Screening
6. Anticipated requirement for surgery or initiation of anti-cancer therapy, other than described in this study protocol, during the study period
7. Known hypersensitivity to any of the combination partners of ATX-101
8. Any malignancy over the last 5 years, other than ovarian/fallopian tube/primary peritoneal cancer, with exception of basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that is considered cured by excision
9. Cardiac failure NYHA III/IV.
10. LVEF < 50% (ECHO or MUGA must not be older than 12 weeks)
11. QTcF > 470 msec
12. Any organ dysfunction or current acute or chronic disease, other than the study indication, that would significantly increase the expected risk in participants participating in the study, in the judgment of the Investigator
13. Pregnant or breast-feeding women
14. Unwilling or unable to follow protocol requirements
15. A past positive status of HIV and/or positive for HIV at Screening
16. Active Hepatitis B or C. In participants with a history of Hepatitis B or Hepatitis C infection, HBsAg and HCV RNA tests have to be negative.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Part 1: To determine the maximum tolerated dose (MTD) of ATX-101 in combination with carboplatin/pegylated liposomal doxorubicin. Measured by incidence of Dose Limiting Toxicity. | Assessed from the time of the first administered dose of ATX-101 up to the last treatment in Cycle 2 (i.e. Days 2 to 30).
  Measured by incidence of Dose Limiting Toxicity (DLT): the MTD is defined as the highest dose level at which ≤ 1/6 of treated participants experience a DLT during a DLT period of 30 days. The RP2D will be either the MTD or the highest tested dose level if MTD is not reached.
Part 2: To assess the progression free survival (PFS) of ATX-101 in combination with carboplatin/pegylated liposomal doxorubicin. Measured by Tumor assessments. | Assessed from Day 1 to Week 85
  Measured by tumor imaging (CT-scan or MRI) in accordance to Response Evaluation Criteria in Solid Tumors (RECIST) every 3 months over a treatment/observation period of 21 months for the individual patient. Tumor images will be compared and changes will be noted over the entire time. PFS means that the sum of diameters of target lesions will not increase by more than 20%, taking as reference the smallest sum measured.

SECONDARY OUTCOMES:
Part 1: To assess the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of ATX-101 in combination with carboplatin/pegylated liposomal doxorubicin. | Assessed from Day 1 to Week 85
  This is a composite outcome measure. Measured by Incidence, severity, and duration of treatment-emergent adverse events (TEAEs) and treatment-related TEAEs according to CTCAE v5.
Part 1: To characterize the plasma PK profile of ATX-101 following IV infusion in combination with carboplatin/pegylated liposomal doxorubicin. | From pre-dose [within 30 min prior to infusion] until 60 min post infusion
  Measured by characterizing the PK profile by estimating the Area under the drug concentration-time curve from time 0 to infinity (AUC0-inf).
Part 2: To assess the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of ATX-101 in combination with carboplatin/pegylated liposomal doxorubicin. | Assessed from Day 1 to Week 85
  This is a composite outcome measure. Measured by Incidence, severity, and duration of treatment-emergent adverse events (TEAEs) and treatment-related TEAEs according to CTCAE v5.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Meniawy, A/Prof, Principal Investigator — Medical Oncologist, Sir Charles Gairdner Hospital Ground Floor, B Block, Hospital Avenue, Nedlands, WA 6009, Australia
Locations (6):
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Peninsula and Southeast Oncology, Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Hospital, Subiaco, Western Australia

IPD SHARING:
Plan to Share IPD: No